CLINICAL TRIAL: NCT06250673
Title: The Effect of the Mediterranean Diet and Low Cholesterol Diet on Serum Lipid Levels in Individuals Receiving Isotretinoin Treatment
Brief Title: Effect of Different Diets on Isotretinoin Users to Serum Lipid Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Collaborators: Okan University (Other)
Responsible Party: Principal Investigator, Umut Uyar, Principal Investigator, Igdir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UUyar1
Record Dates: First submitted 2023-11-23; First posted 2024-02-09 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-02

CONDITIONS: Acne Cystic; Diet, Healthy
Keywords: Mediternian Diet Low Cholesterol Diet Isotretinoin

STUDY DESIGN:
Intervention Model Description: A total of 46 people, 16-16-14.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mediterranean Diet Group (Experimental): Patients taking medication will be given a diet in accordance with the basic Mediterranean diet rules.
  Interventions: Dietary Supplement: Diet experiment
- Low Cholesterol Group (Experimental): Patients taking medication will be given a diet containing <200 mg of cholesterol per day, based on personal wishes.
  Interventions: Dietary Supplement: Diet experiment
- Control Group (No Intervention): They will not take a diet, and take only the medication.

INTERVENTIONS:
Dietary Supplement: Diet experiment — For the isotretinoin users
  Arms: Low Cholesterol Group; Mediterranean Diet Group

SUMMARY:
This research was planned to prevent secondary hyperlipidemia, which may occur due to isotretinoin used in the treatment of severe acne, with diet. There will be three different groups and followed for 12 weeks. Groups will be; Mediterranean Diet, Low Cholesterol Diet (<200 mg/day) and the Control Group.

DETAILED DESCRIPTION:
Isotretinoin has been officially used to treat severe cystic acne since the 1980s. The drug is a retinoic acid derivative and works by reducing the size of the sebaceous glands and sebum production. Thanks to this effect, the lipid profile on the skin surface changes and the bacterial skin flora decreases.

The drug also has a side effect of increasing blood lipids, causing secondary hyperlipidemia. This research examines the effects of low cholesterol diet and Mediterranean diet on blood lipids, which are implemented to prevent the increase of blood lipids.

The research was designed as an experimental intervention research and will conducted at Nevruz Erez State Hospital Skin and Venereology Polyclinics between November 2023 and April 2024, with volunteers who meet the research criteria.

H0: Secondary hyperlipidemia due to isotretinoin use cannot be prevented by diet.

H1: Secondary hyperlipidemia due to isotretinoin use can be prevented by diet. People who volunteer to participate in the research will be informed in detail about the research with the Informed Consent Form and then will be grouped by the list method. At the beginning of the research, the Personal Information Form, the Mediterranean Diet Adherence Scale and the Food Consumption Frequency form prepared by the researcher will be applied to all patients who volunteer to participate in the research. The results of Biochemistry and Hemogram tests performed by the doctor will be recorded.

During the research, the blood findings (Total Cholesterol, HDL-Cholesterol, LDL-Cholesterol, Triglyceride, ALT, AST and Hemogram) of the patients in each group will be checked monthly by the Skin and Venereology Polyclinic Physician who follows their treatment, and the patients' isotretinoin doses will be completely adjusted by the doctor. No intervention other than diet will be made by the researcher.

Sample size of the study (n); Effect size (d) = 0.94, significance level (α) = 0.05, power of the test (1-β) = 80% were entered into the Gpower program and calculated as 32(n) for two groups. This research will be conducted with three different groups, in this case, it is planned to complete the research on a total of at least 48 patients, namely the Mediterranean Diet Group (n1) = 16, the Low Cholesterol Diet Group (n2) = 16 and the Control Group (n3) = 16.

Considering that the research period is 12 weeks, 25% more people will be recruited for each group in case the patients leave the study or are excluded from the research. In this situation; Mediterranean Diet Group (n1) = 20 people, Low Cholesterol Diet Group (n2) = 20 people, Control Group (n3) = 20 people, Total Sample Size (n) = 60 people. The total research duration for all groups participating in the research is planned to be 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients must be treated for acne and must be new to oral isotretinoin treatment, Aged must be 18 - 65 years old, Body Mass Index must be between 18-24.99 kg/m2, LDL Cholesterol must be <130 mg/dL, Triglyceride must be <150 mg/dL.

Exclusion Criteria:

Cardiovascular diseases, Kidney diseases, Eating disorders, Hyperlipidemia, Insulin resistance, Metabolic diseases, Diabetes, And who used the drugs for the treatment of these diseases, BMI <18 kg/m2, >25 kg/m2 Aged <18 and >65 will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Biochemical Tests | 4 weeks, 8 weeks, 12 weeks
  Participants ' blood lipids will be monitored since the research aims to prevent seconder hyperlipidemia. HDL, LDL, Total Cholesterol, Triglyceride, ALT and AST values will be checked monthly.
Mediterranean Diet Adherence Scale | 4 weeks, 8 weeks, 12 weeks
  Within the scope of the research, data will be evaluated with the Mediterranean Diet Adherence Scale, Food Consumption Frequency, Personal Information-Check Form and patients' biochemical test results.
  The validity and reliability study of the Mediterranean Diet Adherence Scale was conducted for Turkey in 2020 by Pehlivanoğlu et al. The scale consists of 14 questions and the answers to these questions are scored between 0 and 1 by the researcher. If the total score obtained from the scale is ≤5, it means low compliance with the Mediterranean diet, if it is between 6-9 points, it means medium compliance with the Mediterranean diet, and if the score is ≥10, it means high compliance with the Mediterranean diet.

SECONDARY OUTCOMES:
Food Consumption Frequency Form | 4 weeks, 8 weeks, 12 weeks
  Within the scope of the research, data will be evaluated with the Mediterranean Diet Adherence Scale, Food Consumption Frequency, Personal Information-Check Form and patients' biochemical test results.
  With the help of the Food Consumption Frequency Form which was created by the researcher, patients' compliance with their diet and how much cholesterol and fat they consume will be checked and recorded monthly.

OTHER OUTCOMES:
Personal Information-Check Form | 4 weeks, 8 weeks, 12 weeks
  With this form, the meal frequencies, medication doses, and physical activities of the participants will be recorded for later use in comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Uyar, Study Director — Igdir University
Locations (1):
- Iğdır Dr. Nevruz Erez State Hospital, Iğdır, Merkez, Turkey (Türkiye)